CLINICAL TRIAL: NCT01083251
Title: The Beneficial Effect of Vitamin D Supplement to Peg Interferon Alpha 2a or to Telbivudine Monotherapy in Patients With Chronic HBV Viral Infection
Brief Title: The Beneficial Effect of Vitamin D Supplement to Peg Interferon Alpha 2a or to Telbivudine Monotherapy in Patients With Chronic Hepatitis B Virus (HBV) Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Assy Nimer, Ziv medical center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 004-10
Record Dates: First submitted 2010-03-03; First posted 2010-03-09 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2010-03

CONDITIONS: Hepatitis B Virus
Keywords: HBV; VITAMIN D; PEGITERFERON; Telbivudine
MeSH Terms: conditions — Hepatitis B | interventions — Vitamin D; Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Peg + Vitamin D (Experimental): Treatment arm with vitamin D will be treated first with vitamin D supplement for 3 months before the initiation of antiviral therapy. Vitamin D levels will be measures at baseline and three months after. The serum vitamin D-25-OH levels should be > 32 ng/ml before the initiation of antiviral treatment). HBV DNA levels will be also measure at baseline and after 3 months of mono therapy with vitamin D
  Interventions: Drug: Peginterferon + Vitamin D
- Peginterferon (Active Comparator)
  Interventions: Drug: Peginterferon
- Sebivo (Active Comparator): Nucleotide Analog Telbivudine 600 mg daily
  Interventions: Drug: Sebivo
- entecavir + vitamin d (Active Comparator): baraclude 1 mg x1/ day + vitamin d
  Interventions: Drug: entecavir+ vitamin d

INTERVENTIONS:
Drug: Peginterferon + Vitamin D — 180 mcg/week + 400 IUX2/day
  Arms: Peg + Vitamin D
Drug: Peginterferon — 180 mcg/week
  Arms: Peginterferon
Drug: Sebivo — Telbivudine 600 mg daily
  Arms: Sebivo
Drug: entecavir+ vitamin d — entecavir 1 mg daily+ vitamin d
  Arms: entecavir + vitamin d

SUMMARY:
Abstract

Telbivudine is a potent inhibitor of HBV but, due to a low genetic barrier to resistance, a high incidence of resistance has been observed in patients with high baseline levels of replication and in those with detectable HBV DNA after 24 weeks of therapy (A1). Telbivudine might be used in patients with good predictors of response (HBV DNA <2 X 106 IU/ ml, i.e. approximately 107 copies/ ml, or 6.3 log 10 IU/ ml at baseline) with verification of HBV DNA suppression below detection in real time PCR assay at 24 weeks.(EASL Guidelines for HBV 2009) The therapy of Pegylated-interferon-alpha-2a is considered as the standard of care for patients with chronic hepatitis b viral infection. However, recent study by Buster et al showed that a sustained viral response (SVR less than 2000 iu.ml at 6 months after treatment)) is obtained in 8 % of patients with genotype D, 30% genotype A, and 20-25% genotypes B or C (47). Vitamin D is a potent immune-modulator; and has been shown to improve SVR in combination with peg interferone in patients with chronic HCV viral infection (48). The impact of vitamin D on virologic response rates of interferon-based treatment of CHB is unknown. The aim of this study therefore was to assess whether Vitamin D, added to the conventional peg therapy in CHB, or to nucleotide analogues could improve the treatment efficacy

ELIGIBILITY:
Inclusion Criteria:

* patients were eligible if they had been HBsAg positive for at least 6 months,
* patients were HBeAg positive or negative,
* patients had increased serum ALT levels between 1 and 10 times the upper limit of normal (ULN),
* patients had serum HBV-DNA levels greater than 1.0 x 10E5 copies/mL (2.0 X 10E4 IUmL), and
* patients had findings on a liver biopsy within the preceding 12 months that were consistent with the presence of chronic hepatitis B.

Exclusion Criteria:

* decompensated liver disease,
* antiviral therapy within 6 months before randomization,
* viral co-infections (hepatitis C virus, hepatitis delta virus, or human immunodeficiency virus), or
* pre-existent neutropenia or thrombocytopenia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
treatment efficacy | 120 weeks
  The primary end point will be sustained viral response which was deﬁned as clearance of HBeAg from serum and HBV DNA less than 10,000 copies/mL (2000 IU/mL) at 6 months after treatment. HBsAg titre during treatment and at 6 months follow up will be measured also (ROCH or Abott Kit).
histologic response | 120 WEEKS
  Another primary endpoint will be histologic response (reduction of at least two points without fibrosis worsening in the total score on the Histological Activity Index).

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Liver clinic, Safed
  - Ziv medical center liver unit, Safed, Israel